CLINICAL TRIAL: NCT05411328
Title: Efficacy of Virtual Reality on Balance in Children With Ataxic Cerebral Palsy Randomized Controlled Trail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, walaa eldesoukey heneidy, lecturer of physical therapy, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: virtual reality and ataxic cp
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Ataxic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy, Ataxic, Autosomal Recessive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional physical therapy group (Experimental): received traditional physical therapy protocol
  Interventions: Device: virtual reality
- virtual reality group (Experimental): received the same traditional physical therapy in addition to virtual reality games
  Interventions: Device: virtual reality

INTERVENTIONS:
Device: virtual reality — All children in the two groups received physical therapy protocol for 30 minutes in addition to virtual reality game traditional physical therapy group traditional physical therapy group

SUMMARY:
Ataxic CP is one type of cerebral palsy. children with ataxic cerebral palsy have trouble with balance and coordination. They may walk with their legs farther apart than other kids and have a hard time with activities that use small hand movements, like writing. Some also have trouble with depth perception This means being able to accurately judge how close or far away something is

ELIGIBILITY:
Inclusion Criteria:

* ataxic cerebral palsy aged 9-14 years

Exclusion Criteria:

* any musculoskeletal conditions that affect balance previous surgeries that affecting balance

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in overall stability index | [Time Frame: baseline and after 3 months of intervention.]
  change in overall stability index will measured by using biodex balance system

CONTACTS AND LOCATIONS:
Locations (1):
- Delta University for Science and Technology, Gamasa, Dakahelia, Egypt

IPD SHARING:
Plan to Share IPD: Yes